CLINICAL TRIAL: NCT06645457
Title: The Effect of Stress Ball and 4-7-8 Breathing Technique on Pre-Procedure Fear, Anxiety and Physiological Parameters in Elderly Patients Undergoing Endoscopy: Randomized Controlled Study
Brief Title: The Effect of Stress Ball and 4-7-8 Breathing Technique on Fear, Anxiety and Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Ayse Gul Parlak, Assistant professor, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KAU-SBF-AGP-03
Record Dates: First submitted 2024-07-02; First posted 2024-10-16 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Endoscopy; Breathing Exercises; Cognitive Therapy; Stress; Anxiety; Physiological Parameters
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- stress ball (Experimental): group applying the stress ball for 20 minute before endoscopy
  Interventions: Other: stress ball
- 4-7-8 breathing technique (Experimental): group applying the 4-7-8 breathing technique for 6 sets before endoscopy
  Interventions: Other: 4-7-8 breathing technique
- Control group (No Intervention): The group in which no intervention was performed before endoscopy and routine care was given

INTERVENTIONS:
Other: stress ball — Patients squeeze the stress ball
  Arms: stress ball
Other: 4-7-8 breathing technique — breathing in quietly through the nose for 4 seconds. holding the breath for a count of 7 seconds. exhaling forcefully through the mouth for 8 seconds.
  Arms: 4-7-8 breathing technique

SUMMARY:
The study aimed to examine the effects of two different applications (stress ball and 4-7-8 breathing technique) before Upper GI Endoscopy on patients' fear, anxiety and physiological parameters before the procedure.

The study as a single-blind, pre-test and post-test experimental study.

DETAILED DESCRIPTION:
Due to the procedures involved, endoscopy patients experience high levels of fear and anxiety. Fear and anxiety may activate the patient's autonomic nervous system, causing increased sweating, heart rate, blood pressure and respiratory rate, and complications related to the procedure. Reducing fear and anxiety and making the patient feel relaxed not only prevents possible harm to the patient due to the procedure, but also facilitates the work of the healthcare team performing the procedure and ensures accurate results. In this context, this study aimed to examine the effects of stress ball exercise and 4-7-8 breathing technique on the fear, anxiety and vital signs of patients who will undergo Upper Gastrointestinal (GI) endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Upper GI Endoscopy will be performed for the first time,
2. American Society of Anesthesiologists (ASA) Status I-II
3. Those over 18 years of age
4. Participates in the research voluntarily and is willing to cooperate.
5. No visual impairment, hearing impairment or communication problem,
6. Not having a psychiatric diagnosis and not using anxiolytic, hypnotic or sedative drugs

Exclusion Criteria:

1. Those diagnosed with severe respiratory failure
2. Those who have health problems in the hand, wrist or arm area that prevent squeezing the stress ball.
3. Using psychiatric medication (antipsychotic, antidepressant, anxiolytic, sedative, etc.
4. Anyone who wishes to leave the research at any stage of the research, with his or her own initiative.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | At the beginning and end of the 20-minute stress ball or breathing exercise intervention (before the endoscopy procedure)
  Developed by Price et al. (1983), VAS is a reliable, valid and practical measurement tool for repeated measurements. The scale, which is generally used to score pain, will be used in this study to score patients' fear between 1-10 points. The scale is represented by a 10 cm line representing the lowest and highest scores for fear (0 = no fear, 10 = most intense fear).
State-Trait Anxiety İnventory | At the beginning and end of the 20-minute stress ball or breathing exercise intervention (before the endoscopy procedure)
  It was developed by Spielberger and his colleagues in 1970. It has two parts: State and Trait Anxiety. The State Anxiety Scale section determines how a person feels at a particular moment and under certain conditions. The feelings or behaviors expressed by the person are answered by marking one of the options: (1) not at all, (2) a little, (3) a lot, (4) completely, depending on the degree of severity. Trait Anxiety Scale is related to how the individual feels in general, regardless of the current situation.

SECONDARY OUTCOMES:
systolic blood pressure (mm/Hg) | At the beginning and end of the 20-minute stress ball or breathing exercise intervention (before the endoscopy procedure)
  Measurements are made at the beginning and end of the stress ball or breathing exercise intervention applied before the endoscopy (before the endoscopy procedure).
diastolic blood pressure (mm/Hg) | At the beginning and end of the 20-minute stress ball or breathing exercise intervention (before the endoscopy procedure)
  Measurement are made at the beginning and end of the stress ball or breathing exercise intervention applied before the endoscopy (before the endoscopy procedure).
SpO2-peripheral oxygen saturation (%) | At the beginning and end of the 20-minute stress ball or breathing exercise intervention (before the endoscopy procedure)
  Measurement are made at the beginning and end of the stress ball or breathing exercise intervention applied before the endoscopy (before the endoscopy procedure).
Respiratory rate (minute value) | At the beginning and end of the 20-minute stress ball or breathing exercise intervention (before the endoscopy procedure)
  Measurement are made at the beginning and end of the stress ball or breathing exercise intervention applied before the endoscopy (before the endoscopy procedure).
heart rate (minute value) | At the beginning and end of the 20-minute stress ball or breathing exercise intervention (before the endoscopy procedure)
  Measurement are made at the beginning and end of the stress ball or breathing exercise intervention applied before the endoscopy (before the endoscopy procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Gül Parlak, PhD, Principal Investigator — Kafkas Üniversity; Mehtap Çullu, PhD, Study Chair — Muğla Üniversity; Zeliha Özkaraca, MSc, Study Chair — muğla provincial directorate of national education
Locations (1):
- Mehtap ÇULLU, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No